CLINICAL TRIAL: NCT00127322
Title: The Early High Risk Period for Patients With Incident Heart Failure: A Population Based Study
Brief Title: The Early High Risk Period for Patients With Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Other Study IDs: 2003EP005B; PG/03/097
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2006-02-13 (Estimated); Status verified 2006-02

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, Congestive; survival; patient admission
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Many people with heart failure either die or are admitted to the hospital in the first few months after the condition is diagnosed. The reasons for this are currently unclear- but may be due to worsening heart failure or other medical conditions such as angina, heart attack or sudden electrical problems of the heart. The investigators propose to recruit and follow-up 450 people, with a new diagnosis of heart failure for a minimum of six months in a multi-centre observational study at two hospital sites: The Hillingdon (Uxbridge) and The Conquest (Hastings) hospitals. The total study duration will be two years. People will be recruited after a diagnosis of heart failure is made and the study will assess reasons for death or admission to hospital and the psychological impact of the condition on both patients and their carers. This is an observational study and no change will be made to patients' conventional treatment.

Hypotheses:

1. The high mortality and hospitalisation rate in the early period after diagnosis of heart failure is related to progressive pump failure; or
2. The high mortality in the early period after the diagnosis of heart failure is related to co-morbid events- principally major coronary events such as myocardial infarction or acute coronary syndrome.

This research should help to identify ways of improving the outlook for people with newly diagnosed heart failure. The analysis of the data generated by this study will be supervised by a statistician. Clinical and demographic data will be described using mean + standard deviation, for continuous variables, and absolute numbers and percentages for categorical variables. Group differences will be examined by t-tests for continuous variables and Chi-square (x2) test for categorical variables. Survival will be reported in terms of Kaplan-Meier curves with differences analysed by Cox proportional hazards.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure

Exclusion Criteria:

* Under age of 18 years
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2004-01; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Cowie, MD MRCP MSc, Principal Investigator — Imperial College London and Royal Brompton NHS Trust; Paresh A Mehta, MBChB MRCP, Principal Investigator — Imperial College and Royal Brompton Trust; Simon W Dubrey, MD MRCP, Principal Investigator — The Hillingdon Hospitals NHS Foundation Trust; Hugh F McIntyre, MD FRCP, Principal Investigator — East Sussex Hospitals NHS Trust; David M Walker, MD FRCP, Principal Investigator — East Sussex Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - The Conquest Hospital, Hastings
  - Hillingdon Hospital, Pield Heath Road, London